CLINICAL TRIAL: NCT06412328
Title: The Effect of Psychosocial Support-based Psychoeducation Program on Psychiatric Symptoms, Stress Coping Styles and Social Support Perceptions of Families of Children and Adolescents Diagnosed with Duchenne Muscular Dystrophy
Brief Title: Psychoeducation Program for Parents of Children with Duchenne Muscular Dystrophy
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: Lokman Hekim University (Other Government)
Responsible Party: Principal Investigator, Başak Çağla Arslan, Lecturer, Lokman Hekim University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 2023109
Record Dates: First submitted 2024-05-07; First posted 2024-05-14 (Actual); Last update posted 2025-03-28 (Actual); Status verified 2025-03

CONDITIONS: Psychoeducation; Parents; Psychological Wellness; Duchenne Muscular Dystrophy
MeSH Terms: conditions — Psychological Well-Being; Muscular Dystrophy, Duchenne

STUDY DESIGN:
Intervention Model Description: Pre-test - post-test, parallel, randomized controlled
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Control group (No Intervention): The parents in the control group did not receive any psychoeducation program
- Intervention group (Experimental): The parents in the intervention group received an 8-session psychoeducation program
  Interventions: Other: Psychoeducation

INTERVENTIONS:
Other: Psychoeducation — The psychoeducation program based on psychosocial support is a total of 8 sessions. Families participating in the study received the psychoeducation program over 4 weeks, with two sessions per week, each session lasting 60 minutes. Parents were included in group work during the psychoeducation program.
  Arms: Intervention group

SUMMARY:
Having and caring for a child with disabilities brings emotional, social and economic difficulties for many families. Families may experience many physiological and psychological problems due to the stress and anxiety they experience. In addition, it is seen that families with children with disabilities give up their existing roles, reduce their participation in social activities, and reach stagnation in their social lives. Mothers are affected psychologically more than fathers and feel lonely. It is stated that mothers believe that they cannot afford everything in the face of the responsibilities they carry and accordingly, they experience emotional and psychological problems such as stress, anxiety, depression, absent-mindedness, forgetfulness and tantrums.

Living with a child with a disability causes family members to experience different emotions as mentioned above; families may frequently experience fear, anxiety, guilt, anger and depression. It is reported that mothers of children with DMD experience depression, anxiety about the future and uncertainty more than mothers of healthy children. Families of children with DMD reported that they felt tired and fatigued during the process of caring for the child and had difficulties in participating in social activities and allocating time for themselves. Most of these families stated that they needed psychological and social support. Therefore, it is important to address the psychiatric aspects of families with children with DMD during the disease process. Parental health contributes positively to the health and adaptation of the family in general. Examining the psychiatric symptoms caused by the problems experienced by families related to DMD and how they cope with this stress will be useful in evaluating and addressing these families. In addition, the social support that families with children with disabilities receive from their immediate environment and institutions is also an important issue. It has been reported that social support from relatives, friends, neighbors, organizations and communities increases the psychological resilience levels of families, they feel that they are not alone in the face of problems, and their anxiety levels decrease. In the literature, it is generally mentioned that when the culture of pediatric care is supportive and family-oriented, the care of the patient will undergo a change when transitioning from pediatric care to the adult period. However, studies evaluating the problems experienced by families in the care of patients with DMD, psychiatric symptoms, ways of coping with stress and perceived social support are insufficient. It is important to evaluate the problems experienced by parents in the families of children with DMD in developing skills to cope with the disease process and disease-related problems, and then to provide training in these areas. Because if parents, who are in the role of caregivers, are equipped with knowledge and skills in this context, they will provide better care and be more useful to their children with DMD.

In line with this information, the aim of this study was to evaluate the problems experienced by parents of children with DMD, psychiatric symptoms, coping skills with stress and the level of social support they perceive and to implement a psychosocial support-based psychoeducation program related to these areas.

ELIGIBILITY:
Inclusion Criteria:

* Having a child diagnosed with DMD
* Volunteering to participate in the study and reading and signing the informed consent form

Exclusion Criteria:

* Having previously or currently participated in any psychoeducation program

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 26 (Estimated)
Dates: Start 2023-06-21 (Actual); Primary Completion 2024-08-29 (Actual); Study Completion 2026-02-28 (Estimated)

PRIMARY OUTCOMES:
Demographic information form | pre-intervention
Brief Symptom Inventory | pre-intervention and immediately after the intervention
  It consists of five sub-dimensions (anxiety, depression, negative self, somatization and hostility) and 53 items. A high score in each sub-dimension indicates an increased level of discomfort in the person.
Coping with stress scale | pre-intervention and immediately after the intervention
  The scale has five sub-dimensions: "self-confident approach", "optimistic approach", "helpless approach", "submissive approach" and "social support seeking approach". The scale consists of 30 items in total and is scored between 0-3. Each sub-dimension is scored separately. In the evaluation of the scale, an increase in the scores obtained from self-confident, optimistic and social support seeking approach means that effective stress coping methods are used, while an increase in the scores of helpless and submissive approach means that ineffective stress coping methods are used.
Multidimensional Scale of Perceived Social Support MSPSS | pre-intervention and immediately after the intervention
  The scale consists of 12 items in total and has three sub-dimensions: "family support, friend support and special person support". The lowest score that can be obtained from the subscales is 4 and the highest score is 28. The lowest score that can be obtained as a total scale score is 12 and the highest score is 84. A high score obtained from the scale means that the perceived social support is also high.

CONTACTS AND LOCATIONS:
Locations (1):
- Lokman Hekim Universiyt, Ankara, Cankaya, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
The results of the study will be published in an article, but participants' information will be kept confidential. It will not be shared with other researchers.